CLINICAL TRIAL: NCT01527084
Title: Timing of Surgical Intervention After Percutaneous Catheter Drainage in STEP UP Approach for Severe Acute Pancreatitis: a Randomized Controlled Stud
Brief Title: Timing of Surgical Intervention After Percutaneous Catheter Drainage in STEP UP Approach for Severe Acute Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajesh Gupta, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8760PG11
Record Dates: First submitted 2012-01-21; First posted 2012-02-06 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): undergo surgery between days 10 - 15 after PCD
  Interventions: Procedure: surgical intervention after percutaneous catheter drainage
- Group B (Other): continued with PCD beyond 15 days and indications for surgery in them will be,
  1. Persistent sepsis or symptoms
  2. Worsening of clinical condition
  3. Failure to thrive
  4. Complications of SAP or PCD
  Interventions: Procedure: surgical intervention after percutaneous catheter drainage

INTERVENTIONS:
Procedure: surgical intervention after percutaneous catheter drainage — Patients who are not improving by day 10 after PCD insertion will be included in the present study and are randomized to group A (early surgery i.e. between 10-15days after PCD insertion ) or group B (Extended treatment with PCD with saline irrigation for more than 15days after PCD insertion)

SUMMARY:
1. To determine the appropriate timing of surgical intervention after Percutaneous Catheter Drainage (PCD) in infected pancreatic necrosis (IPN).
2. To see the change in morbidity and mortality after changing the interval of surgery after PCD

DETAILED DESCRIPTION:
In present study we plan to determine the appropriate timing of surgical intervention after PCD in step up approach of Infected pancreatic necrosis (IPN).

The investigators also intend to evaluate the role of PCD in obviating the surgical intervention in the management of IPN and evaluate the risks & benefits of extended treatment policy of PCD in step up approach of IPN in comparison to early surgery after PCD.

ELIGIBILITY:
Inclusion Criteria:

* All patients with diagnosis of IPN (UK GUIDELINES) managed with percutaneous catheter drainage (PCD) for 10 to 15 days and not showing significant improvement on PCD will be included

Exclusion Criteria:

1. Patient showing significant improvement on PCD within 10 days of its insertion.(Significant improvement on PCD is defined as resolution of fever, acceptance of enteral nutrition, decrease in total leukocyte count, reversal of organ system failure)
2. Sterile pancreatic necrosis
3. An acute intra abdominal event ( perforation of hollow viscus, bleeding, or the abdominal compartment syndrome) during or within 10 days after PCD insertion
4. Previous drainage or surgical necrosectomy for infected pancreatic necrosis (ERCP with or without papillotomy is allowed.)
5. Previous exploratory laparotomy for acute abdomen and diagnosis of pancreatitis during laparotomy

Ages: 14 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mortality | participants will be followed for the duration of hospital stay, an expected average duration of 5 weeks
Reversal of existing organ failure | participants will be followed for the duration of hospital stay, an expected average duration of 5 weeks
New onset multiorgan failure or sepsis and systemic complications | participants will be followed for the duration of hospital stay, an expected average duration of 5 weeks
Locoregional complications | participants will be followed for the duration of hospital stay, an expected average duration of 5 weeks
  Pseudocyst, Pancreatic fistula, Enteric fistula, Perforation of a hollow viscus, and bleeding requiring intervention

SECONDARY OUTCOMES:
Proportion of patients in which surgery would be avoided in Group B | participants will be followed for the duration of hospital stay, an expected average duration of 5 weeks
Pancreatic insufficiency (New onset Diabetes and steatorrhea) | participants will be followed for the duration of hospital discharge to end of our study period, an expected average duration of 1 year
Total number of PCD catheters and catheter related interventions required, and catheter and drain related complications | participants will be followed for the duration of hospital stay, an expected average duration of 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Gupta, MBBS,MS, MCh, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (2):
- India (2):
  - PGIMER, Chandigarh, Chandigarh
  - Postgraduate Institute of Medical Education and Research, Chandigarh